CLINICAL TRIAL: NCT07042217
Title: A Randomized, Double-blind, Parallel-arm, Sham-controlled Trial of ElectraRx Mindfulness Transcranial Direct Current Treatment System (Elect-MDS) for Adults With Major Depressive Disorder
Brief Title: Transcranial Direct Current Stimulation for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soterix Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELECTMDS
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Unipolar Depression
Keywords: tDCS; mindulness; tES; electrotherapy; depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS and Mindfulness (Experimental): Application of electrical stimulation to the brain non-invasively combined with mindfulness
  Interventions: Device: transcranial direct current stimulation (tDCS) and mindfulness instruction
- Sham tDCS and Mindfulness (Sham Comparator): Sham electrical stimulation and mindfulness
  Interventions: Device: Sham tDCS and Mindfulness

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) and mindfulness instruction — tDCS together with audio providing mindfulness instruction and music
  Arms: Active tDCS and Mindfulness
Device: Sham tDCS and Mindfulness — Placebo electrical sitmulation and audio-guided mindfulness instruction
  Arms: Sham tDCS and Mindfulness

SUMMARY:
This study will test the efficacy of transcranial direct current stimulation (tDCS) combined with mindfulness, remotely-delivered using a telemedicine protocol in 25 adults with unipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients that meet criteria for diagnosis of MDD according to DSM-V-TR and confirmed with the Mini International Neuropsychiatric interview
* Currently experiencing a major depressive episode of at least 4 week's duration as part of a unipolar depression
* QIDS-SR score >11 on all three days of screening week (Days 1,3, 7)
* Scored at least 17 (inclusive) on the HDRS-17 at trial entry
* Any antidepressant medication is stable ≥ 30 days prior to HDRS-17 screening
* Female patients are allowed if not pregnant and using a medically acceptable method of contraception, if of childbearing potential.

Exclusion Criteria:

* Failure to respond to at least 2 antidepressant medications
* Drug or alcohol abuse or dependence in the preceding 3 months
* Concurrent benzodiazepine medication
* High suicide risk assessed during clinician screening at baseline interview.
* Failure to respond to ECT treatment or rTMS treatment in this or any previous episode.
* Current DSM-V-TR psychotic disorder
* History of clinically defined neurological disorder or insult that may impact participation in this study as determined by study physician
* Metal in the cranium or skull defects
* Implanted pump, neurostimulator, cardiac pacemaker or defibrillator
* Skin lesions on scalp at the proposed electrode sites
* Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Week 4 and Week 7
  Change in HDRS score from Baseline
Blinding Integrity | Week 7
  Participants will be asked to guess whether they received active or sham treatment, providing a third option of "don't know"

SECONDARY OUTCOMES:
Response and Remission rates defined by HDRS | Week4, Week 7, Week 10, and Week 13
  Response rate, defined as a reduction in the HDRS score by 50% or more, and the remission rate, defined as an HDRS score ≤7.
Quick Inventory of Depressive Symptomatology- Self Report (QIDS-SR) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, and Week 13
  Safety outcome will be tested using the QIDS-SR through a web portal
Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, and Week 13
  Participants will enter responses to the Q-LES-Q-SF questionnaire through the web interface
Clinical Global Impression severity (CGI-S) and improvement (CGI-I) subscales | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, and Week 13
  Participants will enter responses to the CGI-S and CGI-I questionnaires through the web interface
Sheehan Disability Scale (SDS) | Baseline, Week 7, and Week 13
  Participants will be scored on the SDS at Baseline and at the end of the acute and maintenance phases.
Montgomery-Asburg Depression Rating Scale (MADRS) | Baseline, Week 7 and Week 13
  Trained clinical MADRS scores will be obtained at the end of the Acute phase and Maintenance phase.

OTHER OUTCOMES:
Adverse Event Questionnaire | 5 times per week for 7 weeks
  Participants will report any side effects experienced, their severity (mild, moderate, severe), pain scores based on the Wong-Baker pain scale, and temporal relationship with the tDCS session (before, during, after)
Current Mood Score | 5 times per week for 7 weeks
  Participants will enter a daily mood score on a scale of 0-10 (0= feeling normal and not depressed at all and 10= feeling as depressed as they possibly could be) on the web interface

CONTACTS AND LOCATIONS:
Locations (1):
- Soterix Medical, Inc., Woodbridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: Sponsor's webpage with information about the study — https://soterixmedical.com/depression/clinicaltrial